CLINICAL TRIAL: NCT04268511
Title: Ultrasound-Guided Low-dose Caudal Epidural Block Versus Ultrasound-Guided Pudendal Nerve Block for Pediatric Circumcision: A Prospective Observational Study
Brief Title: Caudal Epidural Block Versus Ultrasound-Guided Pudendal Nerve Block for Pediatric Circumcision
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Volkan Ozen, MD, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 1374
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Circumcision
Keywords: Ultrasound; Pudendal nerve block; Caudal epidural block; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caudal epidural block group: Linear ultrasound probe and the sacral hiatus at the sacral cornu level was visualized using an out-of-plane transverse view at 5-10 megahertz . The linear probe was then rotated 90 degrees and placed longitudinally in the midline to evaluate the sacral cornus, sacrococcygeal ligament and sacral bone.
  Interventions: Procedure: Caudal epidural block group
- Pudendal nerve block group: The long axis of the ultrasound probe was positioned on a horizontal line connecting the ischial tuberosity that had been previously located by palpation to the anus. The ischial tuberosity could be easily identified as a hypoechoic area that is bounded superiorly by a hyperechoic line. The probe was then moved medially on the same axis until the rectum appeared as another hypoechoic area.
  Interventions: Procedure: Pudendal nerve block group

INTERVENTIONS:
Procedure: Caudal epidural block group — The linear probe of ultrasound was then rotated 90 degrees and placed longitudinally in the midline to evaluate the sacral cornus, sacrococcygeal ligament and sacral bone. A 22 Gauge 50 mm echogenic block needle was advanced
  Groups: Caudal epidural block group
Procedure: Pudendal nerve block group — A 22 Gauge 50 mm insulated needle was then introduced in the anterior-posterior direction at the middle of the ultrasound probe's superior edge with an out-of-plane approach and using an inclination of 15° in the sagittal plane. The needle tip's position was identified by direct visualization using the movement of adjacent anatomical structures.
  Groups: Pudendal nerve block group

SUMMARY:
The regional anesthesia methods of caudal epidural block (CEB) and dorsal penile nerve block (DPNB) play an important role in providing postoperative pain control in pediatric circumcision surgery. However, the short-term postoperative analgesic effect and the risk of block failure limit the use of DPNB, a peripheral nerve block.

DETAILED DESCRIPTION:
CEB is a neuraxial block and commonly used to control moderate and severe postoperative pain following surgery related to the lumbosacral and midthoracic dermatomes. CEB can have serious undesirable complications such as intravascular and subarachnoid injection, urinary retention and motor block. Pudendal nerve block can be used as an alternative to both DPNB and CEB for penile surgery such as circumcision. The pudendal nerve is a peripheral nerve combining the anterior rami of the sacral plexus nerves (S2-S4) and provides motor and sensory innervation to the perineal region.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged between 4-12 years
* ASA (American Society of Anesthesiologists) I-II group
* Scheduled for circumcision
* Able to communicate in Turkish
* Willing to participate to the study (parents and children)

Exclusion Criteria:

* Patients aged less than 4 or more than 12 years
* Neurological deficit
* Bleeding diathesis
* History of local anesthetic allergy
* Current infection or redness in the region to be injected
* Congenital lower back anomaly
* Liver disease
* Psychiatric disorder
* Mental retardation
* Communication problem
* Refusal to participate in the study.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male patients aged between 4-12 years in the ASA (American Society of Anesthesiologists) I-II group and scheduled for circumcision
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Time of Postoperative analgesic requirement | Up to 12 hours
  It was assessed five times after the operation with Children's Hospital Eastern Ontario Pain Scale. The lowest scale score is 4 points and the highest 13 points. Significant pain behavior for Children's Hospital Eastern Ontario Pain Scale has been identified as 7 points or more. Following transfer from the recovery unit to the ward, the 30 minutes, 1st, 2nd, 6th, and 12th hour pain levels were evaluated by the ward nurse.
Level of Postoperative pain | Up to 12 hours
  It was assessed five times after the operation with Children's Hospital Eastern Ontario Pain Scale. The lowest scale score is 4 points and the highest 13 points. Significant pain behavior for Children's Hospital Eastern Ontario Pain Scale has been identified as 7 points or more. Following transfer from the recovery unit to the ward, the 30 minutes, 1st, 2nd, 6th, and 12th hour pain levels were evaluated by the ward nurse.
Level of Postoperative pain | At the 24th hour
  It was assessed one time for 24th hour by parents with Faces Pain Scale-Revised. The scale is scored in even numbers from 0 to 10, which themselves indicate no pain and significant pain, respectively. The parents were also informed that a scale score of 4 or more

SECONDARY OUTCOMES:
Rate of Postoperative complications | Up to 12 hours
  Urinary retention, nausea, vomiting, lower extremity numbness, motor block were postoperative complications. They were assessed by ward nurse.
Level of Parent satisfaction | Up to 24 hours
  The parents were asked about their satisfaction with the child's comfort and activity level [1, unsatisfied; 2, satisfied (good); 3, absolutely satisfied (excellent)] at the 24-hour follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Ozen, MD, Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Okmeydani Training and Research Hospital, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tutuncu AC, Kendigelen P, Ashyyeralyeva G, Altintas F, Emre S, Ozcan R, Kaya G. Pudendal Nerve Block Versus Penile Nerve Block in Children Undergoing Circumcision. Urol J. 2018 May 3;15(3):109-115. doi: 10.22037/uj.v0i0.4292. PMID 29299888
- [Background] Gaudet-Ferrand I, De La Arena P, Bringuier S, Raux O, Hertz L, Kalfa N, Sola C, Dadure C. Ultrasound-guided pudendal nerve block in children: A new technique of ultrasound-guided transperineal approach. Paediatr Anaesth. 2018 Jan;28(1):53-58. doi: 10.1111/pan.13286. Epub 2017 Dec 5. PMID 29205687
- [Background] Kendigelen P, Tutuncu AC, Emre S, Altindas F, Kaya G. Pudendal Versus Caudal Block in Children Undergoing Hypospadias Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):610-5. doi: 10.1097/AAP.0000000000000447. PMID 27501015